CLINICAL TRIAL: NCT03261037
Title: An International Study to Characterize the Disease Behaviour of Idiopathic Pulmonary Fibrosis and Interstitial Lung Disease During the Peri-Diagnostic Period
Brief Title: A Study to Characterize the Disease Behavior of Idiopathic Pulmonary Fibrosis (IPF) and Interstitial Lung Disease (ILD) During the Peri-Diagnostic Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MA39297; 2016-005114-22 (EudraCT Number)
Record Dates: First submitted 2017-08-22; First posted 2017-08-24 (Actual); Results first posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Idiopathic Pulmonary Fibrosis; Interstitial Lung Disease
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Lung Diseases, Interstitial | interventions — Accelerometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants With Suspicion of IPF/ILD (Other): A participant will be eligible for inclusion if the Investigator has a suspicion that the participant may have IPF/ILD based on symptoms and radiological evidence.
  Interventions: Other: Spirometry; Other: Accelerometry; Other: 6MWT

INTERVENTIONS:
Other: Spirometry — Daily spirometry will be conducted by the participant at home using the study kit provided. Spirometry assessments (FVC) will be conducted at approximately the same time each day with the participant in a seated position. Additionally, site spirometry will also be performed during pre-diagnosis assessment period, on the day of diagnosis, post-diagnosis assessment period, and at end of study.
Other: Accelerometry — Daily physical functional capacity assessments (e.g., steps per day, calorie expenditure) will be measured on an ongoing basis using the accelerometry device provided.
Other: 6MWT — The 6MWT will be performed only at sites where a formalized process is available and the test can be performed under safe conditions, during pre-diagnosis assessment period, on the day of diagnosis, post-diagnosis assessment period, and at end of study.

SUMMARY:
This international clinical study will enroll participants with a suspected diagnosis of IPF/ILD. This study will characterize the disease behavior of IPF and ILD in the peri-diagnostic period. This objective will be achieved using a multidimensional approach assessing changes in pulmonary function, measured by daily handheld spirometry and site spirometry as well as assessing physical functional capacity at home (accelerometry) and at site (6-minute walk tests [6MWT]). Daily handheld spirometry or physical functional capacity assessments are not routinely performed in this participant population. By following participants' lung function before and after diagnosis using home spirometry, levels of physical activity, as well as self-assessment data from the participants (patient reported outcomes; PRO), the study would provide potentially more rapid information on disease behavior and eventually progression compared to usual clinic measurements that occur only every 3-6 months. By receiving data from daily handheld spirometry measurements, treating physicians may have an improved chance of detecting earlier and outside of hospital visits a decline in lung function that could potentially lead to improvements in both diagnosis and treatment for participants with IPF/ILD.

ELIGIBILITY:
Inclusion Criteria:

* Able to comply with the study protocol, in the Investigator's judgment - for example, the ability to use the provided spirometer and tablet and the ability to fill in the required patient reported outcomes questionnaires
* Suspicion of IPF/ILD: radiological evidence of IPF/ILD in symptomatic participants (unexplained dyspnea on exertion and/or cough)

Exclusion Criteria:

* Participation in any investigational study within 28 days prior to inclusion
* History of clinically significant cardiac disease that could explain the patient's symptomatology in the opinion of the Investigator
* Known history of any connective tissue disease, including, but not limited to, rheumatoid arthritis, scleroderma, systemic lupus erythematosus, or mixed connective tissue disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2017-12-25 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (37):
- Canada (4):
  - St. Clare'S Mercy Hospital, St. John's, Newfoundland and Labrador
  - Kingston Health Sciences Centre; research Kingston General Health Research Institute, Kingston, Ontario
  - Dr. Syed Anees Medicine Profession Corporation, Windsor, Ontario
  - Clinique de pneumologie et du sommeil de Lanaudiere, Saint-Charles-Borromée, Quebec
- France (9):
  - Hopital Louis Pradel; Pneumologie, Bron
  - Hopital Cote De Nacre; Pneumologie, Caen
  - Ch De Granville; Pneumologie, Granville
  - Hopital Calmette; Pneumologie, Lille
  - Hopital Arnaud De Villeneuve; Pneumologie A, Montpellier
  - Hopital Tenon;Pneumologie, Paris
  - Centre Pneumologie Et Allergie, Perpignan
  - Hopital de Pontchaillou; Service de Pneumologie, Rennes
  - Ch Bretagne Atlantique; Pneumologie-Oncologie, Vannes
- Ireland (2):
  - Cork University Hospital, Cork
  - St James's Hospital, Dublin
- Italy (12):
  - P.O. Clinicizz. 'SS. Annunziata'; U.O.C. Pneumologia, Chieti, Abruzzo
  - Azienda Ospedaliera dei Colli - P. Monaldi; Dip. Medicina Clinica e Chirurgia, Napoli, Campania
  - A.O. Universitaria Policlinico Di Modena; DIP. Malattie Dell'apparato Respiratorio, Modena, Emilia-Romagna
  - Policlinico A. Gemelli e C.I.C.; Polo Scienze Cardiovascolari e Toraciche - UOC Pneumologia, Rome, Lazio
  - Az. Osp.Univ.San Martino; Pneumologia, Genoa, Liguria
  - ASST Rhodense; U.O.C. Pneumologia, Garbagnate Milanese (MI), Lombardy
  - Ospedale Policlinico S. Matteo; S.C. Pneumologia, Pavia, Lombardy
  - A.O.U. S. Luigi Gonzaga; Interstiziopatie Malattie Rare Polmone, Orbassano (TO), Piedmont
  - A.O.U. Sassari; Dip. Medicina Clinica e Sperimentale, Sassari, Sardinia
  - Az. Osp. Univ. P. Giaccone; UOC di Pneumologia, Palermo, Sicily
  - Pres. Osp. Unico ZT9 - Ospedale Generale Provinciale; U.O.C. Pneumologia, Macerata, The Marches
  - Azienda Ospedaliero-Universitaria Careggi; SOD Pneumologia e Fisiopatologia Toracico Polmonare, Florence, Tuscany
- Netherlands (3):
  - Admiraal de Ruijter Ziekenhuis, Goes
  - Erasmus Medisch Centrum, Rotterdam
  - Isala, Zwolle
- Russia (7):
  - Pulmonologii NII FMBA of Russia, Moscow, Moscow Oblast
  - SBI at Rostov Region "Regional Clinical Hospital #2", Rostov-on-Don, Rostov Oblast
  - SBEI HPE "The First St.Petersburg State Medical University n.a. acad. I.P.Pavlova"of MoH of RF, Saint Petersburg, Sankt-Peterburg
  - SBIH "Chelyabinsk Regional Clinical Hospital", Chelyabinsk, Sverdlovsk Oblast
  - Municipal Healthcare Institution City Clinical Hospital #3 named after M.A. Podgorbunskogo, Kemerovo
  - SBIH at Vladimir Region "Regional Clinical Hospital", Vladimir
  - Budget Institution of Healthcare of Voronezh Region "Voronezh Regional Clinical Hospital #1", Voronezh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wijsenbeek MS, Bendstrup E, Valenzuela C, Henry MT, Moor CC, Jouneau S, Fois AG, Moran-Mendoza O, Anees S, Mirt M, Bengus M, Gilberg F, Kirchgaessler KU, Vancheri C. Disease Behaviour During the Peri-Diagnostic Period in Patients with Suspected Interstitial Lung Disease: The STARLINER Study. Adv Ther. 2021 Jul;38(7):4040-4056. doi: 10.1007/s12325-021-01790-y. Epub 2021 Jun 11. PMID 34117601
- [Derived] Wijsenbeek M, Bendstrup E, Valenzuela C, Henry MT, Moor C, Bengus M, Perjesi A, Gilberg F, Kirchgaessler KU, Vancheri C. Design of a Study Assessing Disease Behaviour During the Peri-Diagnostic Period in Patients with Interstitial Lung Disease: The STARLINER Study. Adv Ther. 2019 Jan;36(1):232-243. doi: 10.1007/s12325-018-0845-3. Epub 2018 Nov 30. PMID 30506309

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled participants in Canada, France, Ireland, Italy, the Netherlands, and Russia.
Groups:
- IPF Participants: Participants diagnosed with Idiopathic Pulmonary Fibrosis (IPF)
- Non-IPF ILD Participants: Participants diagnosed with an Interstitial Lung Disease (ILD) other than Idiopathic Pulmonary Fibrosis (non-IPF)
- Non-ILD Participants: Participants diagnosed with a condition that was not an Interstitial Lung Disease (non-ILD)
- Participants Without Diagnosis: Participants without diagnosis
Period: Overall Study
Arm/Group | IPF Participants | Non-IPF ILD Participants | Non-ILD Participants | Participants Without Diagnosis
Started | 68 | 62 | 9 | 39
Completed | 64 | 41 | 9 | 11
Not Completed | 4 | 21 | 0 | 28
Not completed — Withdrawal by Subject | 2 | 13 | 0 | 18
Not completed — Non-compliance with study procedures | 0 | 2 | 0 | 6
Not completed — Participant moving away and can no longer be in study | 0 | 1 | 0 | 0
Not completed — Participant came out of study due to investigator discretion | 0 | 2 | 0 | 0
Not completed — Diagnosed but protocol deviation | 1 | 0 | 0 | 0
Not completed — Participant did not want to continue the study | 0 | 1 | 0 | 0
Not completed — Participant did not want to continue the diagnostic procedures | 0 | 0 | 0 | 1
Not completed — Participant presented clinical improvement | 0 | 2 | 0 | 0
Not completed — Technical difficulties | 0 | 0 | 0 | 1
Not completed — Equipment failed to work | 0 | 0 | 0 | 1
Not completed — End of study for participant and no follow up | 0 | 0 | 0 | 1
Not completed — Participant was too weak to continue in study | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IPF Participants | Non-IPF ILD Participants | Non-ILD Participants | Participants Without Diagnosis | Total
Number analyzed (Participants) | 68 | 62 | 9 | 39 | 178
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.3 (6.97) | 65.1 (9.99) | 69.6 (7.7) | 71.2 (8.64) | 68.3 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 32 | 3 | 12 | 66
  Male | 49 | 30 | 6 | 27 | 112
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaskan Native | 1 | 0 | 0 | 0 | 1
  White | 62 | 50 | 7 | 24 | 143
  Unknown | 0 | 1 | 0 | 0 | 1
  Missing | 5 | 11 | 2 | 15 | 33
Race/Ethnicity, Customized [Number; unit: Participant]
  Hispanic or Latino | 9 | 12 | 0 | 1 | 22
  Not Hispanic or Latin | 49 | 36 | 7 | 20 | 112
  Not reported | 4 | 3 | 0 | 2 | 9
  Unknown | 1 | 0 | 0 | 1 | 2
  Missing | 5 | 11 | 2 | 15 | 33

OUTCOME MEASURES:

1. Primary Outcome: Time-Adjusted Semi-Annual Forced Vital Capacity (FVC) Decline in Participants With IPF During the Peri-Diagnostic Period, Measured in Milliliters (mL) by Daily Home Spirometry
Description: Minimum site visits were: baseline, diagnosis, and EOS for each participant. From inclusion into the study, participants were followed for up to12 months. The EOS was defined as: If no diagnosis was made 12 months after inclusion, the participant left the study; Participants diagnosed with non-ILD left the study on the date of diagnosis; Participants diagnosed with IPF or non-IPF ILD were followed up to the start of drug treatment (within 6 months) or up to 6 months if no drug treatment was prescribed. Therefore, the total length of the study was variable for each participant. Measurements were taken daily by home spirometry. The semi-annual mean FVC decline was calculated by use of the estimated semi-annual FVC decline of each individual participant. The individual FVC decline was estimated by applying a linear regression model to all acceptable FVC measurements flagged as 'Good blow' collected by the individual participant during the entire peri-diagnostic period (up to 18 months).
Time Frame: From Day 1 into the study to end of the study (up to 18 months) and adjusted for 6 months. There was no fixed visit schedule for the whole study and reported results comprise all data points from enrollment to EOS
Population: Participants diagnosed with IPF. Only participants for whom data were collected are included in the analysis.
Measure: Mean (Standard Deviation); unit: milliliter (mL)
Arm/Group | IPF Participants
Number analyzed (Participants) | 64
milliliter (mL) | -308.7 (1268.72)

2. Secondary Outcome: Time-Adjusted Semi-Annual FVC Decline in Participants With Non-IPF ILD During the Peri-Diagnostic Period, Measured in mL by Daily Home Spirometry
Description: as for outcome 1
Time Frame: as for outcome 1
Population: Participants diagnosed with non-IPF ILD. Only participants for whom data were collected are included in the analysis.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Non-IPF ILD Participants
Number analyzed (Participants) | 59
mL | 57.5 (1277.03)

3. Secondary Outcome: Change From Baseline in the FVC Decline in IPF and Non-IPF ILD Participants During the Peri-Diagnostic Period, Measured in mL by Site Spirometry
Description: The peri-diagnostic period covered the pre-diagnostic period (from inclusion into the study (enrollment visit), participants were followed for a maximum of 12 months in the pre-diagnostic assessment period) and the post-diagnostic period (from diagnosis to the start of drug treatment within 6 months or a maximum of 6 months if no drug treatment was prescribed).
Time Frame: From Baseline to end of the study (up to 18 months)
Population: Participants diagnosed with IPF and non-IPF ILD. Only participants for whom data were collected are included in the analysis.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | IPF Participants | Non-IPF ILD Participants
Number analyzed (Participants) | 68 | 62
mL
  Baseline: number analyzed (Participants) | 66 | 61
  Baseline | 2845.6 (814.83) | 2782.4 (870.24)
  Change from Baseline at End of Study Visit: number analyzed (Participants) | 62 | 59
  Change from Baseline at End of Study Visit | -51.3 (270.56) | -27.1 (265.52)

4. Secondary Outcome: Change From Baseline in the Percent Predicted FVC in IPF and Non-IPF ILD Participants During the Peri-Diagnostic Period, Measured by Site Spirometry
Description: as for outcome 3
Time Frame: From Baseline to end of the study (up to 18 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent Predicted (%)
Arm/Group | IPF Participants | Non-IPF ILD Participants
Number analyzed (Participants) | 68 | 62
Percent Predicted (%)
  Baseline: number analyzed (Participants) | 66 | 61
  Baseline | 82.8 (18.74) | 83.9 (17.82)
  Change form Baseline at End of Study Visit: number analyzed (Participants) | 62 | 59
  Change form Baseline at End of Study Visit | -0.6 (7.26) | -0.6 (8.49)

5. Secondary Outcome: Change From Baseline in Distance Walked (Meters) on the 6MWT in IPF and Non-IPF ILD Participants During the Peri-Diagnostic Period, Assessed at Site
Description: The 6MWT measures the distance a patient is able to walk quickly on a flat, hard surface in a period of 6 minutes. The peri-diagnostic period covered the pre-diagnostic period (from inclusion into the study (enrollment visit), participants were followed for a maximum of 12 months in the pre-diagnostic assessment period) and the post-diagnostic period (from diagnosis to the start of drug treatment within 6 months or a maximum of 6 months if no drug treatment was prescribed).
Time Frame: From Baseline to end of the study (up to 18 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Meter (m)
Arm/Group | IPF Participants | Non-IPF ILD Participants
Number analyzed (Participants) | 68 | 62
Meter (m)
  Baseline: number analyzed (Participants) | 66 | 60
  Baseline | 434.6 (117.30) | 429.4 (139.51)
  Change from Baseline at End of Study Visit: number analyzed (Participants) | 63 | 55
  Change from Baseline at End of Study Visit | 4.4 (96.18) | 6.4 (87.97)

6. Secondary Outcome: Decline in Physical Function Capacity (Steps/Day) in IPF and Non-IPF ILD Participants During the Peri-Diagnostic Period, Measured by Daily Home Accelerometry
Description: Patients were asked to wear an accelerometer during the course of the study which provided information on their physical activity at home, with daily measurements used to investigate the development of physical function capacity. The peri-diagnostic period covered the pre-diagnostic period (from inclusion into the study (enrollment visit), participants were followed for a maximum of 12 months in the pre-diagnostic assessment period) and the post-diagnostic period (from diagnosis to the start of drug treatment within 6 months or a maximum of 6 months if no drug treatment was prescribed).
Time Frame: From inclusion into the study to end of the study (up to 18 months)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Steps per Day
Arm/Group | IPF Participants | Non-IPF ILD Participants
Number analyzed (Participants) | 66 | 61
Steps per Day | -1237.2 (14146.07) | -13407.3 (72612.82)

7. Secondary Outcome: Calorie Expenditure in IPF and Non-IPF ILD Participants During the Peri-Diagnostic Period, Measured by Daily Home Accelerometry
Time Frame: From inclusion into the study to end of the study (up to 18 months)
Population: Data collection was impacted by technical problems that could not be solved, thus invalid data collected was not analyzed.
Measure: Number; unit: Calorie
Arm/Group | IPF Participants | Non-IPF ILD Participants
Number analyzed (Participants) | 68 | 62
Calorie | NA — Calorie expenditure device was malfunctioning and unreliable data were collected, which was not suitable to analyse therefore there was no analysis done. | NA — Calorie expenditure device was malfunctioning and unreliable data were collected, which was not suitable to analyse therefore there was no analysis done.

8. Secondary Outcome: Change in the King's Brief Interstitial Lung Disease (K-BILD) Questionnaire Total Score by Visit During the Peri-Diagnostic Period
Description: The K-BILD questionnaire was specifically developed to analyze the health status of participants with ILD. The questionnaire consists of 15 items (assessed by the patients on a scale ranging from 1 to 7, where 1 and 7 represent worst and best health status). Items are compiled into 3 domains: breathlessness and activities (range: 0-21), psychological (range: 0-34) , and chest symptoms (range: 0-8). To score the K-BILD, the Likert response scale weightings for individual items are combined and scores are transformed to a range of 0-100 by using logit values (higher scores indicate better health status). The peri-diagnostic period covered the pre-diagnostic period (from enrollment visit participants were followed for up to 12 months) and the post-diagnostic period (from diagnosis to the start of drug treatment within 6 months or a maximum of 6 months if no drug treatment was prescribed).
Time Frame: From inclusion into the study to end of the study (up to 18 months)
Population: All enrolled participants completed the questionnaire. Only participants for whom data were collected are included in the analysis.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | IPF Participants | Non-IPF ILD Participants | Non-ILD Participants | Participants Without Diagnosis
Number analyzed (Participants) | 68 | 62 | 9 | 39
Units on scale
  Baseline: number analyzed (Participants) | 68 | 62 | 9 | 38
  Baseline | 60.57 (17.633) | 55.70 (14.203) | 54.22 (11.703) | 60.47 (15.728)
  Change from Baseline at End of Study Visit: number analyzed (Participants) | 63 | 60 | 9 | 24
  Change from Baseline at End of Study Visit | -0.45 (9.709) | 3.98 (11.851) | 6.03 (14.294) | 4.01 (9.313)

9. Secondary Outcome: Modified Medical Research Council (mMRC) Dyspnea Scale Scores During the Peri-Diagnostic Period
Description: The mMRC dyspnea scale was used to grade the effects of breathlessness on daily activities over time. The following grading categories are used for this scale: Grade 0 - I only get breathless with strenuous exercise; Grade 1 - I get short of breath when hurrying on the level or walking up a slight hill; Grade 2 - I walk slower than people of the same age on the level because of breathlessness or have to stop for breath when walking on my own pace; Grade 3 - I stop for breath after walking about 100 yards or after a few minutes on level ground; Grade 4 - I am too breathless to leave the house. The peri-diagnostic period covered the pre-diagnostic period (from inclusion into the study (enrollment visit), participants were followed for a maximum of 12 months in the pre-diagnostic assessment period) and the post-diagnostic period (from diagnosis to the start of drug treatment within 6 months or a maximum of 6 months if no drug treatment was prescribed).
Time Frame: From inclusion into the study to end of the study (up to 18 months)
Population: All enrolled participants. Only participants for whom data were collected are included in the analysis. Data of post-diagnosis period for non-ILD participants and participants without diagnosis were not collected.
Measure: Count of Participants; unit: Participants
Arm/Group | IPF Participants | Non-IPF ILD Participants | Non-ILD Participants | Participants Without Diagnosis
Number analyzed (Participants) | 68 | 61 | 9 | 32
Participants
  Pre-diagnosis: number analyzed (Participants) | 30 | 29 | 7 | 20
  Pre-diagnosis: Grade 0 | 12 | 10 | 2 | 6
  Pre-diagnosis: Grade 1 | 8 | 8 | 1 | 11
  Pre-diagnosis: Grade 2 | 7 | 9 | 3 | 2
  Pre-diagnosis: Grade 3 | 3 | 2 | 1 | 1
  Pre-diagnosis: Grade 4 | 0 | 0 | 0 | 0
  Initial diagnosis: number analyzed (Participants) | 68 | 61 | 8 | 3
  Initial diagnosis: Grade 0 | 22 | 17 | 3 | 2
  Initial diagnosis: Grade 1 | 31 | 25 | 0 | 0
  Initial diagnosis: Grade 2 | 10 | 16 | 3 | 1
  Initial diagnosis: Grade 3 | 5 | 3 | 2 | 0
  Initial diagnosis: Grade 4 | 0 | 0 | 0 | 0
  Post-diagnosis: number analyzed (Participants) | 6 | 3 | 0 | 0
  Post-diagnosis: Grade 0 | 2 | 1 |  |
  Post-diagnosis: Grade 1 | 4 | 2 |  |
  Post-diagnosis: Grade 2 | 0 | 0 |  |
  Post-diagnosis: Grade 3 | 0 | 0 |  |
  Post-diagnosis: Grade 4 | 0 | 0 |  |
  End of Study: number analyzed (Participants) | 65 | 61 | 9 | 32
  End of Study: Grade 0 | 20 | 17 | 3 | 13
  End of Study: Grade 1 | 30 | 25 | 1 | 15
  End of Study: Grade 2 | 10 | 16 | 3 | 3
  End of Study: Grade 3 | 5 | 3 | 2 | 1
  End of Study: Grade 4 | 0 | 0 | 0 | 0

10. Secondary Outcome: The EuroQol 5-Dimension 5-Level Questionnaire (EQ-5D-5L) 5-Item Health State Profile Scores During the Peri-Diagnostic Period
Description: The EQ-5D-5L questionnaire is a self-reported health status questionnaire that assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each item is rated by the participant on a five-point scale indicating the followings: Level 1 - no problem; Level 2 - slight problems; Level 3 - moderate problems; Level 4 - severe problems; Level 5 - extreme problems. The peri-diagnostic period covered the pre-diagnostic period (from inclusion into the study (enrollment visit), participants were followed for a maximum of 12 months in the pre-diagnostic assessment period) and the post-diagnostic period (from diagnosis to the start of drug treatment within 6 months or a maximum of 6 months if no drug treatment was prescribed).
Time Frame: From inclusion into the study to end of the study (up to 18 months)
Population: All enrolled participants. Data of post-diagnosis period for non-ILD participants and participants without diagnosis were not collected as participants already discontinued from the study.
Measure: Count of Participants; unit: Participants
Arm/Group | IPF Participants | Non-IPF ILD Participants | Non-ILD Participants | Participants Without Diagnosis
Number analyzed (Participants) | 68 | 62 | 9 | 38
Participants
  Baseline Mobility: Level 1 | 33 | 25 | 2 | 24
  Baseline Mobility: Level 2 | 16 | 15 | 2 | 9
  Baseline Mobility: Level 3 | 14 | 21 | 5 | 4
  Baseline Mobility: Level 4 | 5 | 1 | 0 | 1
  Baseline Mobility: Level 5 | 0 | 0 | 0 | 0
  Baseline Mobility: Missing | 0 | 0 | 0 | 0
  Baseline Self-care: Level 1 | 55 | 52 | 6 | 34
  Baseline Self-care: Level 2 | 7 | 6 | 2 | 4
  Baseline Self-care: Level 3 | 6 | 4 | 1 | 0
  Baseline Self-care: Level 4 | 0 | 0 | 0 | 0
  Baseline Self-care: Level 5 | 0 | 0 | 0 | 0
  Baseline Self-care: Missing | 0 | 0 | 0 | 0
  Baseline Usual activities: Level 1 | 32 | 29 | 4 | 20
  Baseline Usual activities: Level 2 | 19 | 16 | 2 | 10
  Baseline Usual activities: Level 3 | 16 | 15 | 2 | 4
  Baseline Usual activities: Level 4 | 1 | 2 | 0 | 4
  Baseline Usual activities: Level 5 | 0 | 0 | 1 | 0
  Baseline Usual activities: Missing | 0 | 0 | 0 | 0
  Baseline Pain/Discomfort: Level 1 | 29 | 25 | 3 | 20
  Baseline Pain/Discomfort: Level 2 | 22 | 22 | 2 | 10
  Baseline Pain/Discomfort: Level 3 | 17 | 14 | 3 | 4
  Baseline Pain/Discomfort: Level 4 | 0 | 1 | 1 | 3
  Baseline Pain/Discomfort: Level 5 | 0 | 0 | 0 | 1
  Baseline Pain/Discomfort: Missing | 0 | 0 | 0 | 0
  Baseline Anxiety/Depression: Level 1 | 38 | 24 | 5 | 19
  Baseline Anxiety/Depression: Level 2 | 22 | 20 | 2 | 12
  Baseline Anxiety/Depression: Level 3 | 5 | 15 | 2 | 7
  Baseline Anxiety/Depression: Level 4 | 2 | 2 | 0 | 0
  Baseline Anxiety/Depression: Level 5 | 1 | 1 | 0 | 0
  Baseline Anxiety/Depression: Missing | 0 | 0 | 0 | 0
  Pre-diagnosis Mobility: number analyzed (Participants) | 30 | 29 | 7 | 21
  Pre-diagnosis Mobility: Level 1 | 16 | 11 | 1 | 13
  Pre-diagnosis Mobility: Level 2 | 4 | 9 | 2 | 4
  Pre-diagnosis Mobility: Level 3 | 9 | 5 | 2 | 1
  Pre-diagnosis Mobility: Level 4 | 1 | 3 | 2 | 2
  Pre-diagnosis Mobility: Level 5 | 0 | 0 | 0 | 0
  Pre-diagnosis Mobility: Missing | 0 | 1 | 0 | 1
  Pre-diagnosis Self-care: number analyzed (Participants) | 30 | 29 | 7 | 21
  Pre-diagnosis Self-care: Level 1 | 25 | 25 | 5 | 20
  Pre-diagnosis Self-care: Level 2 | 3 | 2 | 2 | 0
  Pre-diagnosis Self-care: Level 3 | 1 | 1 | 0 | 0
  Pre-diagnosis Self-care: Level 4 | 1 | 0 | 0 | 0
  Pre-diagnosis Self-care: Level 5 | 0 | 0 | 0 | 0
  Pre-diagnosis Self-care: Missing | 0 | 1 | 0 | 1
  Pre-diagnosis Usual activities: number analyzed (Participants) | 30 | 29 | 7 | 21
  Pre-diagnosis Usual activities: Level 1 | 15 | 15 | 2 | 9
  Pre-diagnosis Usual activities: Level 2 | 10 | 6 | 3 | 6
  Pre-diagnosis Usual activities: Level 3 | 4 | 7 | 2 | 4
  Pre-diagnosis Usual activities: Level 4 | 1 | 0 | 0 | 0
  Pre-diagnosis Usual activities: Level 5 | 0 | 0 | 0 | 1
  Pre-diagnosis Usual activities: Missing | 0 | 1 | 0 | 1
  Pre-diagnosis Pain/Discomfort: number analyzed (Participants) | 30 | 29 | 7 | 21
  Pre-diagnosis Pain/Discomfort: Level 1 | 15 | 15 | 1 | 12
  Pre-diagnosis Pain/Discomfort: Level 2 | 11 | 7 | 4 | 3
  Pre-diagnosis Pain/Discomfort: Level 3 | 3 | 5 | 0 | 4
  Pre-diagnosis Pain/Discomfort: Level 4 | 1 | 1 | 2 | 0
  Pre-diagnosis Pain/Discomfort: Level 5 | 0 | 0 | 0 | 1
  Pre-diagnosis Pain/Discomfort: Missing | 0 | 1 | 0 | 1
  Pre-diagnosis Anxiety/Depression: number analyzed (Participants) | 30 | 29 | 7 | 21
  Pre-diagnosis Anxiety/Depression: Level 1 | 14 | 12 | 2 | 10
  Pre-diagnosis Anxiety/Depression: Level 2 | 11 | 10 | 4 | 8
  Pre-diagnosis Anxiety/Depression: Level 3 | 3 | 6 | 1 | 1
  Pre-diagnosis Anxiety/Depression: Level 4 | 0 | 0 | 0 | 0
  Pre-diagnosis Anxiety/Depression: Level 5 | 2 | 0 | 0 | 1
  Pre-diagnosis Anxiety/Depression: Missing | 0 | 1 | 0 | 1
  Initial diagnosis Mobility: number analyzed (Participants) | 68 | 62 | 8 | 3
  Initial diagnosis Mobility: Level 1 | 31 | 26 | 2 | 2
  Initial diagnosis Mobility: Level 2 | 19 | 17 | 3 | 0
  Initial diagnosis Mobility: Level 3 | 12 | 9 | 2 | 0
  Initial diagnosis Mobility: Level 4 | 3 | 6 | 1 | 0
  Initial diagnosis Mobility: Level 5 | 0 | 0 | 0 | 0
  Initial diagnosis Mobility: Missing | 3 | 4 | 0 | 1
  Initial diagnosis Self-care: number analyzed (Participants) | 68 | 62 | 8 | 3
  Initial diagnosis Self-care: Level 1 | 55 | 44 | 6 | 2
  Initial diagnosis Self-care: Level 2 | 3 | 10 | 1 | 0
  Initial diagnosis Self-care: Level 3 | 6 | 4 | 1 | 0
  Initial diagnosis Self-care: Level 4 | 1 | 0 | 0 | 0
  Initial diagnosis Self-care: Level 5 | 0 | 0 | 0 | 0
  Initial diagnosis Self-care: Missing | 3 | 4 | 0 | 1
  Initial diagnosis Usual activities: number analyzed (Participants) | 68 | 62 | 8 | 3
  Initial diagnosis Usual activities: Level 1 | 31 | 27 | 6 | 2
  Initial diagnosis Usual activities: Level 2 | 20 | 14 | 1 | 0
  Initial diagnosis Usual activities: Level 3 | 9 | 14 | 1 | 0
  Initial diagnosis Usual activities: Level 4 | 4 | 3 | 0 | 0
  Initial diagnosis Usual activities: Level 5 | 1 | 0 | 0 | 0
  Initial diagnosis Usual activities: Missing | 3 | 4 | 0 | 1
  Initial diagnosis Pain/Discomfort: number analyzed (Participants) | 68 | 62 | 8 | 3
  Initial diagnosis Pain/Discomfort: Level 1 | 32 | 34 | 2 | 1
  Initial diagnosis Pain/Discomfort: Level 2 | 22 | 14 | 1 | 1
  Initial diagnosis Pain/Discomfort: Level 3 | 10 | 6 | 3 | 0
  Initial diagnosis Pain/Discomfort: Level 4 | 1 | 4 | 2 | 0
  Initial diagnosis Pain/Discomfort: Level 5 | 0 | 0 | 0 | 0
  Initial diagnosis Pain/Discomfort: Missing | 3 | 4 | 0 | 1
  Initial diagnosis Anxiety/Depression: number analyzed (Participants) | 68 | 62 | 8 | 3
  Initial diagnosis Anxiety/Depression: Level 1 | 30 | 25 | 4 | 1
  Initial diagnosis Anxiety/Depression: Level 2 | 21 | 17 | 1 | 1
  Initial diagnosis Anxiety/Depression: Level 3 | 10 | 13 | 1 | 0
  Initial diagnosis Anxiety/Depression: Level 4 | 2 | 3 | 2 | 0
  Initial diagnosis Anxiety/Depression: Level 5 | 2 | 0 | 0 | 0
  Initial diagnosis Anxiety/Depression: Missing | 3 | 4 | 0 | 1
  Post-diagnosis Mobility: number analyzed (Participants) | 6 | 3 | 0 | 0
  Post-diagnosis Mobility: Level 1 | 2 | 0 |  |
  Post-diagnosis Mobility: Level 2 | 1 | 2 |  |
  Post-diagnosis Mobility: Level 3 | 2 | 1 |  |
  Post-diagnosis Mobility: Level 4 | 0 | 0 |  |
  Post-diagnosis Mobility: Level 5 | 0 | 0 |  |
  Post-diagnosis Mobility: Missing | 1 | 0 |  |
  Post-diagnosis Self-care: number analyzed (Participants) | 6 | 3 | 0 | 0
  Post-diagnosis Self-care: Level 1 | 4 | 2 |  |
  Post-diagnosis Self-care: Level 2 | 0 | 1 |  |
  Post-diagnosis Self-care: Level 3 | 1 | 0 |  |
  Post-diagnosis Self-care: Level 4 | 0 | 0 |  |
  Post-diagnosis Self-care: Level 5 | 0 | 0 |  |
  Post-diagnosis Self-care: Missing | 1 | 0 |  |
  Post-diagnosis Usual activities: number analyzed (Participants) | 6 | 3 | 0 | 0
  Post-diagnosis Usual activities: Level 1 | 2 | 2 |  |
  Post-diagnosis Usual activities: Level 2 | 2 | 0 |  |
  Post-diagnosis Usual activities: Level 3 | 1 | 1 |  |
  Post-diagnosis Usual activities: Level 4 | 0 | 0 |  |
  Post-diagnosis Usual activities: Level 5 | 0 | 0 |  |
  Post-diagnosis Usual activities: Missing | 1 | 0 |  |
  Post-diagnosis Pain/Discomfort: number analyzed (Participants) | 6 | 3 | 0 | 0
  Post-diagnosis Pain/Discomfort: Level 1 | 1 | 2 |  |
  Post-diagnosis Pain/Discomfort: Level 2 | 4 | 0 |  |
  Post-diagnosis Pain/Discomfort: Level 3 | 0 | 1 |  |
  Post-diagnosis Pain/Discomfort: Level 4 | 0 | 0 |  |
  Post-diagnosis Pain/Discomfort: Level 5 | 0 | 0 |  |
  Post-diagnosis Pain/Discomfort: Missing | 1 | 0 |  |
  Post-diagnosis Anxiety/Depression: number analyzed (Participants) | 6 | 3 | 0 | 0
  Post-diagnosis Anxiety/Depression: Level 1 | 3 | 0 |  |
  Post-diagnosis Anxiety/Depression: Level 2 | 1 | 2 |  |
  Post-diagnosis Anxiety/Depression: Level 3 | 1 | 1 |  |
  Post-diagnosis Anxiety/Depression: Level 4 | 0 | 0 |  |
  Post-diagnosis Anxiety/Depression: Level 5 | 0 | 0 |  |
  Post-diagnosis Anxiety/Depression: Missing | 1 | 0 |  |
  End of Study Mobility: number analyzed (Participants) | 65 | 62 | 9 | 33
  End of Study Mobility: Level 1 | 33 | 28 | 2 | 16
  End of Study Mobility: Level 2 | 15 | 15 | 3 | 2
  End of Study Mobility: Level 3 | 11 | 14 | 3 | 4
  End of Study Mobility: Level 4 | 4 | 3 | 1 | 2
  End of Study Mobility: Level 5 | 0 | 0 | 0 | 0
  End of Study Mobility: Missing | 2 | 2 | 0 | 9
  End of Study Self-care: number analyzed (Participants) | 65 | 62 | 9 | 33
  End of Study Self-care: Level 1 | 54 | 46 | 6 | 22
  End of Study Self-care: Level 2 | 3 | 12 | 2 | 1
  End of Study Self-care: Level 3 | 5 | 2 | 1 | 1
  End of Study Self-care: Level 4 | 1 | 0 | 0 | 0
  End of Study Self-care: Level 5 | 0 | 0 | 0 | 0
  End of Study Self-care: Missing | 2 | 2 | 0 | 9
  End of Study Usual activities: number analyzed (Participants) | 65 | 62 | 9 | 33
  End of Study Usual activities: Level 1 | 32 | 25 | 4 | 14
  End of Study Usual activities: Level 2 | 16 | 18 | 0 | 5
  End of Study Usual activities: Level 3 | 11 | 15 | 4 | 4
  End of Study Usual activities: Level 4 | 3 | 2 | 1 | 1
  End of Study Usual activities: Level 5 | 1 | 0 | 0 | 0
  End of Study Usual activities: Missing | 2 | 2 | 0 | 9
  End of Study Pain/Discomfort: number analyzed (Participants) | 65 | 62 | 9 | 33
  End of Study Pain/Discomfort: Level 1 | 30 | 34 | 2 | 14
  End of Study Pain/Discomfort: Level 2 | 20 | 16 | 1 | 3
  End of Study Pain/Discomfort: Level 3 | 13 | 8 | 4 | 6
  End of Study Pain/Discomfort: Level 4 | 0 | 2 | 2 | 1
  End of Study Pain/Discomfort: Level 5 | 0 | 0 | 0 | 0
  End of Study Pain/Discomfort: Missing | 2 | 2 | 0 | 9
  End of Study Anxiety/Depression: number analyzed (Participants) | 65 | 62 | 9 | 33
  End of Study Anxiety/Depression: Level 1 | 28 | 25 | 4 | 13
  End of Study Anxiety/Depression: Level 2 | 21 | 19 | 1 | 10
  End of Study Anxiety/Depression: Level 3 | 10 | 15 | 2 | 0
  End of Study Anxiety/Depression: Level 4 | 2 | 1 | 2 | 1
  End of Study Anxiety/Depression: Level 5 | 2 | 0 | 0 | 0
  End of Study Anxiety/Depression: Missing | 2 | 2 | 0 | 9

11. Secondary Outcome: The EuroQol Visual Analogue Scale (EQ-VAS) Health State Profile Scores During the Peri-Diagnostic Period During the Peri-Diagnostic Period
Description: The EQ-VAS questionnaire is a self-reported questionnaire that measures health state. The VAS is a 100 mm scale from worst (0 mm) to best (100 mm) health the participant can imagine. The peri-diagnostic period covered the pre-diagnostic period (from inclusion into the study (enrollment visit), participants were followed for a maximum of 12 months in the pre-diagnostic assessment period) and the post-diagnostic period (from diagnosis to the start of drug treatment within 6 months or a maximum of 6 months if no drug treatment was prescribed).
Time Frame: From inclusion into the study to end of the study (up to 18 months)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | IPF Participants | Non-IPF ILD Participants | Non-ILD Participants | Participants Without Diagnosis
Number analyzed (Participants) | 68 | 62 | 9 | 39
Scores on a scale
  Health State Index Baseline: number analyzed (Participants) | 68 | 61 | 9 | 38
  Health State Index Baseline | 71.7 (15.96) | 67.4 (20.11) | 68.9 (17.99) | 76.2 (17.09)
  Health State Index Pre-diagnosis: number analyzed (Participants) | 30 | 28 | 7 | 20
  Health State Index Pre-diagnosis | 69.8 (15.50) | 71.5 (15.89) | 65.7 (19.88) | 73.5 (16.06)
  Health State Index Initial diagnosis: number analyzed (Participants) | 65 | 58 | 8 | 2
  Health State Index Initial diagnosis | 69.5 (16.23) | 68.3 (18.03) | 70.4 (19.92) | 72.5 (10.61)
  Health State Index Post-diagnosis: number analyzed (Participants) | 5 | 3 | 0 | 0
  Health State Index Post-diagnosis | 69.0 (25.10) | 76.7 (12.58) |  |
  Health State Index End of Study: number analyzed (Participants) | 63 | 60 | 9 | 24
  Health State Index End of Study | 69.5 (16.46) | 69.8 (17.21) | 67.0 (21.21) | 74.2 (16.85)

12. Secondary Outcome: The EuroQoL 5-dimension 5-level Questionnaire Index Utility Scores During the Peri-Diagnostic Period
Description: The EQ-5D-5L questionnaire is a self-reported health status questionnaire that assesses mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. A unique health state is defined for each participant by combining the levels from each of the 5 dimensions. Each state is referred to in terms of a 5 digit code, e.g. state 11111 indicates no problems on any of the 5 dimensions, while state 12345 indicates no problems with mobility, slight problems with washing or dressing, moderate problems with usual activities, severe pain or discomfort and extreme anxiety or depression. From these 5 answers an index value is derived between 0 and 1, with a higher value corresponding with a better Quality of Life.
Time Frame: From inclusion into the study to end of the study (up to 18 months)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | IPF Participants | Non-IPF ILD Participants | Non-ILD Participants | Participants Without Diagnosis
Number analyzed (Participants) | 68 | 62 | 9 | 39
Scores on a scale
  Index utility score Baseline: number analyzed (Participants) | 68 | 62 | 9 | 38
  Index utility score Baseline | 0.83 (0.140) | 0.79 (0.143) | 0.67 (0.250) | 0.80 (0.187)
  Index utility score Pre-diagnosis: number analyzed (Participants) | 30 | 28 | 7 | 20
  Index utility score Pre-diagnosis | 0.82 (0.154) | 0.80 (0.152) | 0.68 (0.237) | 0.83 (0.182)
  Index utility score Initial diagnosis: number analyzed (Participants) | 65 | 58 | 8 | 2
  Index utility score Initial diagnosis | 0.81 (0.162) | 0.78 (0.197) | 0.63 (0.331) | 0.92 (0.013)
  Index utility score Post-diagnosis: number analyzed (Participants) | 5 | 3 | 0 | 0
  Index utility score Post-diagnosis | 0.81 (0.149) | 0.75 (0.123) |  |
  Index utility score End of Study: number analyzed (Participants) | 63 | 60 | 9 | 24
  Index utility score End of Study | 0.81 (0.164) | 0.80 (0.164) | 0.62 (0.312) | 0.81 (0.197)

13. Secondary Outcome: Fatigue Assessment Scale (FAS) Score During the Peri-Diagnostic Period
Description: The FAS is a fatigue questionnaire consisting of 10 items; five questions reflect physical fatigue and five questions analyze mental fatigue. A five-point scale (one for "never" to five for "always") is used for participant responses. The scale score is calculated by summing all items. Therefore, the FAS scores can range from 10 to 50. The peri-diagnostic period covered the pre-diagnostic period (from inclusion into the study (enrollment visit), participants were followed for a maximum of 12 months in the pre-diagnostic assessment period) and the post-diagnostic period (from diagnosis to the start of drug treatment within 6 months or a maximum of 6 months if no drug treatment was prescribed).
Time Frame: From inclusion into the study to end of the study (up to 18 months)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | IPF Participants | Non-IPF ILD Participants | Non-ILD Participants | Participants Without Diagnosis
Number analyzed (Participants) | 68 | 62 | 9 | 39
Scores on a Scale
  Baseline: number analyzed (Participants) | 67 | 60 | 9 | 37
  Baseline | 21.8 (6.44) | 21.8 (6.89) | 21.1 (7.22) | 20.9 (6.99)
  Initial diagnosis: number analyzed (Participants) | 64 | 56 | 7 | 2
  Initial diagnosis | 21.7 (6.66) | 22.6 (7.33) | 24.7 (9.11) | 18.0 (2.83)
  End of study: number analyzed (Participants) | 63 | 58 | 8 | 24
  End of study | 22.0 (6.17) | 22.0 (7.59) | 26.1 (9.33) | 20.6 (6.31)

14. Secondary Outcome: Cough, Urge to Cough, and Fatigue Visual Analogue Scales (VAS) Score During the Peri-Diagnostic Period
Description: The VAS are 100 mm scales on which participants indicate the severity of their cough, the urge to cough and their fatigue. In the VAS, participants had to record their health state on a scale ranging from 0 (best imaginable health state) to 100 (worst imaginable health state). A mean of this health state was recorded for participant analyzed in this outcome measure. The peri-diagnostic period covered the pre-diagnostic period (from inclusion into the study (enrollment visit), participants were followed for a maximum of 12 months in the pre-diagnostic assessment period) and the post-diagnostic period (from diagnosis to the start of drug treatment within 6 months or a maximum of 6 months if no drug treatment was prescribed).
Time Frame: From inclusion into the study to end of the study (up to 18 months)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | IPF Participants | Non-IPF ILD Participants | Non-ILD Participants | Participants Without Diagnosis
Number analyzed (Participants) | 68 | 62 | 9 | 39
Scores on a Scale
  Baseline (Cough): number analyzed (Participants) | 68 | 60 | 9 | 38
  Baseline (Cough) | 34.0 (25.44) | 26.9 (20.66) | 17.9 (21.99) | 27.4 (20.38)
  Pre-diagnosis (Cough): number analyzed (Participants) | 30 | 28 | 7 | 20
  Pre-diagnosis (Cough) | 36.8 (25.50) | 25.4 (20.90) | 11.4 (14.03) | 31.4 (24.34)
  Initial diagnosis (Cough): number analyzed (Participants) | 65 | 58 | 8 | 2
  Initial diagnosis (Cough) | 36.3 (29.60) | 21.9 (18.88) | 17.1 (21.69) | 32.0 (36.77)
  Post-diagnosis (Cough): number analyzed (Participants) | 5 | 3 | 0 | 0
  Post-diagnosis (Cough) | 25.6 (20.94) | 17.0 (9.16) |  |
  End of Study (Cough): number analyzed (Participants) | 63 | 60 | 9 | 24
  End of Study (Cough) | 34.7 (26.64) | 24.0 (19.42) | 19.3 (21.35) | 31.2 (25.92)
  Baseline (Urge to Cough): number analyzed (Participants) | 68 | 60 | 9 | 38
  Baseline (Urge to Cough) | 33.3 (25.41) | 28.6 (21.53) | 16.4 (17.20) | 25.8 (21.27)
  Pre-diagnosis (Urge to Cough): number analyzed (Participants) | 30 | 28 | 7 | 19
  Pre-diagnosis (Urge to Cough) | 37.6 (25.73) | 23.1 (20.03) | 13.2 (13.51) | 30.4 (24.29)
  Initial diagnosis (Urge to Cough): number analyzed (Participants) | 65 | 58 | 8 | 2
  Initial diagnosis (Urge to Cough) | 36.4 (29.22) | 22.9 (19.02) | 13.7 (19.86) | 38.5 (47.38)
  Post-diagnosis (Urge to Cough): number analyzed (Participants) | 5 | 3 | 0 | 0
  Post-diagnosis (Urge to Cough) | 23.5 (15.79) | 10.8 (9.00) |  |
  End of Study (Urge to Cough): number analyzed (Participants) | 63 | 60 | 9 | 23
  End of Study (Urge to Cough) | 33.8 (25.18) | 24.3 (20.14) | 16.2 (20.00) | 36.3 (29.75)
  Baseline (Fatigue): number analyzed (Participants) | 68 | 60 | 9 | 38
  Baseline (Fatigue) | 38.4 (27.15) | 39.4 (24.29) | 30.0 (31.18) | 33.2 (26.89)
  Pre-diagnosis (Fatigue): number analyzed (Participants) | 30 | 28 | 7 | 20
  Pre-diagnosis (Fatigue) | 34.1 (27.50) | 31.0 (22.68) | 32.5 (26.11) | 32.0 (28.29)
  Initial diagnosis (Fatigue): number analyzed (Participants) | 65 | 58 | 8 | 2
  Initial diagnosis (Fatigue) | 37.5 (27.50) | 35.6 (23.79) | 31.1 (30.00) | 17.0 (5.66)
  Post-diagnosis (Fatigue): number analyzed (Participants) | 5 | 3 | 0 | 0
  Post-diagnosis (Fatigue) | 30.4 (23.24) | 25.3 (19.48) |  |
  End of Study (Fatigue): number analyzed (Participants) | 63 | 60 | 9 | 24
  End of Study (Fatigue) | 38.3 (26.15) | 34.6 (23.54) | 35.5 (32.16) | 31.5 (24.18)

15. Secondary Outcome: Pearson's Correlation Coefficient of FVC (mL) Between Home and Site Spirometry in IPF and Non-IPF ILD Participants During the Peri-Diagnostic Period
Description: The correlation of FVC (mL) between home and site spirometry was analyzed by taking into account the individually estimated linear regression models of each participant for home-based FVC measurements and site FVC measurements. This analysis was performed for participants diagnosed with IPF or non-IPF ILD in the peri-diagnosis period. The peri-diagnostic period covered the pre-diagnostic period (from inclusion into the study (enrollment visit), participants were followed for a maximum of 12 months in the pre-diagnostic assessment period) and the post-diagnostic period (from diagnosis to the start of drug treatment within 6 months or a maximum of 6 months if no drug treatment was prescribed).
Time Frame: From inclusion into the study to end of the study (up to 18 months)
Population: Only IPF and non-IPF ILD participants with non-zero declines are included in the analysis.
Measure: Number; unit: Pearson's Correlation Coefficients
Arm/Group | IPF Participants | Non-IPF ILD Participants
Number analyzed (Participants) | 57 | 55
Pearson's Correlation Coefficients | -0.06 | 0.35

16. Secondary Outcome: Pearson's Correlation Coefficient of Physical Functional Capacity Assessed at Home in Terms of the Decline in the Number of Footsteps and on Site in Terms of the Decline in Distance of the 6MWT
Description: The measure represents the correlation of distance walked (meter) assessed by physical function capacity at home and the 6MWT at the site in the peri-diagnosis period. The peri-diagnostic period covered the pre-diagnostic period (from inclusion into the study (enrollment visit), participants were followed for a maximum of 12 months in the pre-diagnostic assessment period) and the post-diagnostic period (from diagnosis to the start of drug treatment within 6 months or a maximum of 6 months if no drug treatment was prescribed).
Time Frame: From inclusion into the study to end of the study (up to 18 months)
Population: Only IPF and non-IPF ILD participants with non-zero declines are included in the analysis.
Measure: Number; unit: Pearson's Correlation Coefficients
Arm/Group | IPF Participants | Non-IPF ILD Participants
Number analyzed (Participants) | 54 | 52
Pearson's Correlation Coefficients | -0.04 | 0.06

17. Secondary Outcome: Percentage of Participants Requiring Respiratory-Related Hospitalizations
Description: The number of participants requiring the hospitalization were counted during pre- and post-diagnosis period.
Time Frame: From inclusion into the study to end of the study (up to 18 months)
Population: All enrolled participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | IPF Participants | Non-IPF ILD Participants | Non-ILD Participants | Participants Without Diagnosis
Number analyzed (Participants) | 68 | 62 | 9 | 39
Percentage of Participants
  With at least one event during pre-diagnosis period | 5.9 | 4.8 | 22.2 | 2.6
  With at least one event during post-diagnosis period | 0 | 0 | 0 | 0

18. Secondary Outcome: Percentage of Participants With Non-Elective Hospitalizations
Description: The number of participants requiring the hospitalization were counted during pre- and post-diagnosis period. Investigator-reported acute exacerbations, deaths, and events related to study assessments were only collected in the clinical database. As the study had no protocol mandated IMP or treatment requirements, any untoward occurrences such as AEs and SAEs were not collected.
Time Frame: From inclusion into the study to end of the study (up to 18 months)
Population: All enrolled participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | IPF Participants | Non-IPF ILD Participants | Non-ILD Participants | Participants Without Diagnosis
Number analyzed (Participants) | 68 | 62 | 9 | 39
Percentage of Participants
  With at least one event during pre-diagnosis period | 8.8 | 4.8 | 22.2 | 7.7
  With at least one event during post-diagnosis period | 2.9 | 0 | 0 | 0

19. Secondary Outcome: Percentage of Participants With Investigator-Reported Acute Exacerbations
Description: Acute exacerbation was defined as per Collard et al. 2016. Investigator-reported acute exacerbations, deaths, and events related to study assessments were only collected in the clinical database. As the study had no protocol mandated IMP or treatment requirements, any untoward occurrences such as AEs and SAEs were not collected.
Time Frame: From inclusion into the study to end of the study (up to 18 months)
Population: All enrolled participants. Data of post-diagnosis period for non-ILD participants and participants without diagnosis were not collected.
Measure: Number; unit: Percentage of Participants
Arm/Group | IPF Participants | Non-IPF ILD Participants | Non-ILD Participants | Participants Without Diagnosis
Number analyzed (Participants) | 62 | 62 | 9 | 39
Percentage of Participants
  With at least one acute exacerbation pre-diagnosis period | 1.5 | 0 | 0 | 0
  With at least one acute exacerbation during post-diagnosis period: number analyzed (Participants) | 62 | 62 | 0 | 0
  With at least one acute exacerbation during post-diagnosis period | 0 | 0 |  |
  With at least one triggered acute exacerbation pre-diagnosis period | 4.4 | 0 | 0 | 0
  With at least one triggered acute exacerbation during post-diagnosis period: number analyzed (Participants) | 62 | 62 | 0 | 0
  With at least one triggered acute exacerbation during post-diagnosis period | 0 | 0 |  |
  With at least one idiopathic acute exacerbation pre-diagnosis period | 0 | 1.6 | 0 | 0
  With at least one idiopathic acute exacerbation during post-diagnosis period: number analyzed (Participants) | 62 | 62 | 0 | 0
  With at least one idiopathic acute exacerbation during post-diagnosis period | 0 | 0 |  |

20. Secondary Outcome: Percentage of Participants Who Died Due to Any Cause
Description: The number of participants, who died due to any cause, were counted during pre- and post-diagnosis period.
Time Frame: From inclusion into the study to end of the study (up to 18 months)
Population: All enrolled participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | IPF Participants | Non-IPF ILD Participants | Non-ILD Participants | Participants Without Diagnosis
Number analyzed (Participants) | 68 | 62 | 9 | 39
Percentage of Participants | 0 | 0 | 0 | 0

21. Secondary Outcome: Percentage of Participants Who Died Due to Respiratory-Related Diseases
Description: The number of participants, who died due to respiratory-related diseases, were counted during pre- and post-diagnosis period.
Time Frame: From inclusion into the study to end of the study (up to 18 months)
Population: All enrolled participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | IPF Participants | Non-IPF ILD Participants | Non-ILD Participants | Participants Without Diagnosis
Number analyzed (Participants) | 68 | 62 | 9 | 39
Percentage of Participants | 0 | 0 | 0 | 0

22. Secondary Outcome: Percentage of Participants With Events Related to the Study Assessments
Description: The number of participants with events related to the study assessments were counted during pre- and post-diagnosis period. Investigator-reported acute exacerbations, deaths, and events related to study assessments were only collected in the clinical database. As the study had no protocol mandated IMP or treatment requirements, any untoward occurrences such as AEs and SAEs were not collected.
Time Frame: From inclusion into the study to end of the study (up to 18 months)
Population: All enrolled participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | IPF Participants | Non-IPF ILD Participants | Non-ILD Participants | Participants Without Diagnosis
Number analyzed (Participants) | 68 | 62 | 9 | 39
Percentage of Participants | 0 | 3.2 | 0 | 5.1

ADVERSE EVENTS:
Time Frame: From inclusion into the study to end of the study (up to 18 months)
Description: The study had no protocol mandated IMP or treatment requirements. Participants stopped the study prior to starting any drug treatment for IPF/ILD. Any untoward occurrences thought to be due to or associated with a commercial medicinal product used during the course of a participant's standard medical treatment were not reported in the clinical database, but should have been reported to the respective Market Authorization Holder/ local Health Authority according to local regulatory requirements.
Groups:
- Participants With and an ILD Other Than IPF (Non-IPF ILD): Participants diagnosed with an Interstitial Lung Disease (ILD) other than Idiopathic Pulmonary Fibrosis (non-IPF)
Arm/Group | IPF Participants | Participants With and an ILD Other Than IPF (Non-IPF ILD) | Non-ILD Participants | Participants Without Diagnosis
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/62 | 0/9 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/37/NCT03261037/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-11): https://cdn.clinicaltrials.gov/large-docs/37/NCT03261037/SAP_001.pdf